CLINICAL TRIAL: NCT03832270
Title: SPARCLAR: A Feasibility Randomised Controlled Trial of a Parenting Support Programme Focussed on Families Affected by ADHD
Brief Title: Support for PARents of Children Living With ADHD - a Research Trial
Acronym: SPARCLAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Collaborators: NHS Fife (Other Government); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Principal Investigator, Lucy Thompson, International Research Coordinator & Research Fellow, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HIPS/17/58
Record Dates: First submitted 2018-12-04; First posted 2019-02-06 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Parenting support
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Parallel pilot RCT (MRC feasibility phase)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and assessors will be blind to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parents InC (Experimental): Group parenting support intervention based around four pillars: 1) empowerment/ownership; 2) education on ADHD and its effect on family identity/ values; 3) positive parenting in the context of ADHD; 4) making sense of ADHD in a developmental context. It is delivered over 5 weekly 2-hour sessions, a 6 week break, and a follow-up session.
  Interventions: Behavioral: Parents InC
- Incredible Years (Active Comparator): A group parenting support intervention aimed at strengthening parent-child interactions and attachment, reducing harsh discipline and fostering parents' ability to promote children's social, emotional, and academic development. The IY programme is delivered over 14 weekly 2-hour sessions. IY facilitators are videotaped during sessions to maintain intervention fidelity. IY also includes 1-4 pre-intervention preparation sessions which may involve home visits and telephone support and reminders.
  Interventions: Behavioral: Incredible Years

INTERVENTIONS:
Behavioral: Parents InC — Based on social learning theory, Parents InC has been designed specifically for parents of children with an ADHD diagnosis with a particular focus on parenting sense of self competence.
  Arms: Parents InC
Behavioral: Incredible Years — Also based on social learning theory but focus is not specifically on ADHD.
  Arms: Incredible Years

SUMMARY:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a chronic and pervasive disorder characterised by problems in attention, impulse control and activity regulation that substantially burdens patients, families, and society. The efficacy of behavioural training for parents of children with ADHD symptoms is well established, however it is less clear which type of parenting intervention should be offered, and which aspects of parenting behaviour to focus on. It is not established whether an intervention designed specifically for families of children with a diagnosis will be more effective and cost effective than less specifically-targeted interventions. The purpose of this study is to determine the feasibility and likely size of a substantive randomised controlled trial comparing an AHDH specific parenting intervention to a diagnostically less-specific parenting intervention.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a chronic and pervasive disorder characterised by problems in attention, impulse control and activity regulation that substantially burdens patients, families, and society. ADHD is often associated with challenging behaviours that can induce negativity, even in parents who would otherwise cope well.The efficacy of behavioural training for parents of children with ADHD symptoms is well established, however it is less clear which type of parenting intervention should be offered, and which aspects of parenting behaviour to focus on. It is not established whether an intervention designed specifically for families of children with a diagnosis will be more effective and cost effective than less specifically-targeted interventions.

Parents In Control (Parents InC) offers specific support around empowerment, information and behaviour management specific to ADHD, as well as understanding of the child's development context. Parents InC has been used for a number of years in Scotland and has been evaluated, with promising results, but with relatively small sample sizes, no long-term follow-up, no economic evaluation and, most crucially, no comparison to an alternative intervention or to a control group. The investigators now need to understand if it: i) is at least as effective as the current best-evidenced alternative, Incredible Years, in impacting children's behaviour outcomes; ii) is cost-effective; and iii) offers something helpful and unique compared to other parenting programmes in terms of parenting self-competence and quality of life.

The purpose of this study is to determine the feasibility and likely size of a substantive randomised controlled trial comparing an ADHD specific parenting intervention to a diagnostically less-specific parenting intervention (Incredible Years). Specific objectives are to test (1) whether parents of children recently diagnosed with ADHD are willing to be randomised to Parents InC or IY; (2) whether sufficient numbers of families can be (a) recruited and (b) retained such that a full-scale RCT is likely to be feasible; (3) whether research procedures and efficacy measures are feasible and acceptable to participating families (including health economic measures and consent to link to routine datasets); (4) whether families participating in Parents InC achieve similar scores on the parenting sense of competence scale at 12 months post randomisation as those in the comparison arm (Incredible Years); (5) Whether the two intervention arms significantly differ on any other measures; and (6) the mean cost per participant of Parents InC.

ELIGIBILITY:
Inclusion Criteria:

• Parents of children aged 5-12 with a formal diagnosis of ADHD, following a standardised assessment from a paediatrician or a psychiatrist, referred to the Fife integrated ADHD pathway during the one year recruitment period will be eligible for inclusion.

Exclusion Criteria:

* Families attending other parenting groups
* Parents who have low proficiency in English (as this will compromise their ability to complete research measures or participate in a group intervention).
* Participants already taking part in research on a parenting intervention will also be ineligible to participate.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Number of parents willing to be randomised to Parents InC or Incredible Years. | Continuous over 1 year study period
  Measured by number of parents agreed to randomisation throughout the study period.
Number of parents recruited and retained. | Continuous over 1 year study period
  Measured by number of parents recruited and retained throughout the study period.
Research procedures feasibility and acceptability | Continuous over 1 year study period
  Face to face interviews will be conducted with participating families to assess the feasibility and acceptability of research procedures.

SECONDARY OUTCOMES:
Primary efficacy outcome: Parental Sense of Competence Scale. | Baseline, 12-months post-randomisation
  17-items measure of parenting self-esteem questionnaire with 2 sub scales. Each item is rated on a 6 point Likert scale anchored by 1= "Strongly Disagree" and 6= "Strongly Agree". A higher score indicates a higher parenting sense of competency. There are no average scores or 'cut-off's' for this tool.
Eyberg Child Behaviour Inventory. | Baseline, 12-month post-randomisation
  36-items measure (parent reported) that assesses the current frequency and severity of child's behaviour. Items are rated on a 7-point intensity scale and a yes/no Problem scale.
General Health Questionnaire. | Baseline, 12-month post-randomisation
  12-items self-report measure of common psychiatric conditions of parents. Each item is accompanied with four responses; "Not at all", "No more than usual", "Rather more than usual" and "Much more than usual". Items are rated on a 4-point response scale.
ADHD Symptom Rating Scale-Version 1. | Baseline, 12-month post-randomisation
  Self-report symptom checklist consisting of 18 DSM-IV criteria for parents. The checklist assesses occurrence frequency of each symptom.
Parenting Daily Hassles Scale. | Baseline, 3 months post Baseline (if applicable), 12-month post-randomisation
  18-items self-report measure of the frequency and intensity of 20 potential parenting 'hassles' to indicate parents stress. The items are rated on a frequency and intensity scale. The frequency scale is scored rarely =1, sometimes= 2, a lot= 3, and constantly = 4. The intensity scale is scored by adding the parents rating of 1-5 for each item. If a 0 has been scored for frequency on an item then it should be scored 0 for intensity. The range for this scale is 0 -100. This measure will be re-collected if there is > 3 months wait period between baseline data collection and the start date of the parenting groups. This will allow the investigators to detect any baseline measure changes over the wait period.
Goal Based Outcomes. | Baseline, 3 months post Baseline (if applicable), 12-month post-randomisation
  Taken from the Child Outcomes Research Consortium to identify goals and assess progression. Progress toward individual goal is rated on a scale from 0 (no progress) to 10 (goal has been reached). This measure will be re-collected if there is > 3 months wait period between baseline data collection and the start date of the parenting groups. This will allow the investigators to detect any baseline measure changes over the wait period.
EQ-5D-5L | Baseline, 3 months post Baseline (if applicable), 12-month post-randomisation
  Self-report measure of parent quality of life. The EQ-5D-5L is a descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, some problems, moderate problems, extreme problems. Parents will be also be asked to rate their health on a visual analogue scale. This measure will be re-collected if there is > 3 months wait period between baseline data collection and the start date of the parenting groups. This will allow the investigators to detect any baseline measure changes over the wait period.
Paediatric Quality of Life Inventory (PedsQL) | Baseline, 12-month post-randomisation
  23-items questionnaire which covers 4 core dimensions (physical, social, emotional and school functioning). Each dimension has 4 levels: never = 0, almost never= 1, sometimes= 2, often= 3 and almost always= 4.
Strengths and Difficulties Questionnaire (SDQ) | Baseline, 3 months post Baseline (if applicable), 12-month post-randomisation
  25-items questionnaire which assesses child's emotional and behavioural problems. Each item is scored 0, 1 or 2. Somewhat true is always scored 1, but whether Not true and Certainly true are scored 0 or 2 depends on whether the item is framed as a strength or difficulty. This measure will be re-collected if there is > 3 months wait period between baseline data collection and the start date of the parenting groups. This will allow the investigators to detect any baseline measure changes over the wait period.
Participant service use | 12-month post-randomisation
  Measured using diaries

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Thompson, Principal Investigator — University of Glasgow; Helen Minnis, Principal Investigator — University of Glasgow
Locations (1):
- NHS Fife Psychology Department, Dunfermline, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The PIs will manage access rights to the data set. We anticipate that anonymised trial data may be shared with other researchers to enable international prospective meta-analyses.

REFERENCES:
- [Derived] Sim F, Dalgarno L, McIntosh E, Haig C, Duklas P, McConnachie A, Gillberg C, Minnis H, Thompson L. Families with neurodevelopmental diagnoses are not 'Hard to Reach': Findings from a feasibility trial comparing parenting programmes for parents of children with ADHD. PLoS One. 2025 Sep 17;20(9):e0323959. doi: 10.1371/journal.pone.0323959. eCollection 2025. PMID 40961127